CLINICAL TRIAL: NCT03600636
Title: Medium-term Follow-up of Patients With Obstetric Antiphospholipid Syndrome: MRI Study of White Matter
Acronym: APS Follow Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LOCAL/2018/JCG-01
Record Dates: First submitted 2018-06-29; First posted 2018-07-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other)
  Interventions: Procedure: Diffusion tensor imaging MRI
- antiphospholipid syndrome patients (Other)
  Interventions: Procedure: Diffusion tensor imaging MRI

INTERVENTIONS:
Procedure: Diffusion tensor imaging MRI — 1. axial diffusion weighted sequence with 32 gradient encoding directions and two values b, 0 s / mm 2 and 1000 s / mm 2.
  2. Fluid-attenuated inversion recovery
  3. three-dimensional axial image weighted in T1
  4. axial echo-planar image sequence
  5. three-dimensional pulse sequence axial flight time

SUMMARY:
The investigators hypothesize that the white matter of patients with obstetric antiphospholipid syndrome deteriorates over time

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* For the target population: only women included in the publication by Pereira et al (2016) will be included, with no obsteric history (fetal death >10 weeks or 3 unexplained consecutive losses <10 weeks)
* For the test group: Patients must be positive for antiphospholipid antibodies based on results from Pereira et al (2016)
* For the control group. Patients must be negative for antiphospholipid antibodies according to results from Pereira et al (2016)

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant, parturient or breast feeding
* The patient is claustrophobic
* The patient has a metallic foreign body (e.g. pacemaker)
* The patient has experienced pregnancy loss linked to infectious, metabolic, anatomic or hormonal factors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Mean diffusivity of white matter between groups | Day 0
  mm2/s

SECONDARY OUTCOMES:
Fractional anisotropy of white matter between groups | Day 0
  Value between 0-1
Radial diffusivity of white matter between groups | Day 0
  mm2/s
Mean diffusivity of white matter between controls vs subgroups with only anticardiolipin or Lupus anticoagulant and/or aβ2GP1 antiphospholipid antibodies | Day 0
  mm2/s
Fractional anisotropy of white matter between controls vs subgroups with only anticardiolipin or Lupus anticoagulant and/or aβ2GP1 antiphospholipid antibodies | Day 0
  Value between 0-1
Radial diffusivity of white matter between controls vs subgroups with only anticardiolipin or Lupus anticoagulant and/or aβ2GP1 antiphospholipid antibodies | Day 0
  mm2/s

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Gris, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Background] Pereira FR, Macri F, Jackowski MP, Kostis WJ, Gris JC, Beregi JP, Mekkaoui C. Diffusion tensor imaging in patients with obstetric antiphospholipid syndrome without neuropsychiatric symptoms. Eur Radiol. 2016 Apr;26(4):959-68. doi: 10.1007/s00330-015-3922-x. Epub 2015 Jul 23. PMID 26201292
- [Result] Gris JC, Chea M, Bouvier S, Pereira FR. Antiphospholipid Antibodies in Mental Disorders. Semin Thromb Hemost. 2025 Jun;51(4):448-456. doi: 10.1055/s-0044-1788696. Epub 2024 Jul 24. PMID 39047993